CLINICAL TRIAL: NCT04065230
Title: A Prospective,Multi-center,Cohort Trial: the Efficacy and Safety of Tenofovir Alafenamide Fumarate Tablets (TAF) in Blocking Mother-to-child Transmission of Hepatitis B Virus(HBV)
Brief Title: Study of Tenofovir Alafenamide Fumarate Tablets (TAF) in Blocking Mother-to-child Transmission of Hepatitis B Virus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Guo-rong Han, Director of Obstetrics and Gynecology, Southeast University, China
Other Study IDs: H201908
Record Dates: First submitted 2019-08-18; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis B Virus; Mother to Child Transmission
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 64 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAF antiviral therapy group
  Interventions: Drug: Tenofovir Alafenamide Fumarate tablets

INTERVENTIONS:
Drug: Tenofovir Alafenamide Fumarate tablets — Eligible hepatitis B pregnant women are given TAF antiviral therapy (25mg, oral, 1/day) at 24-28 weeks of gestation until one month after delivery.

SUMMARY:
This study is a single-group, multi-center and prospective clinical study designed to assess the efficacy and safety of TAF in blocking mother-to-child transmission of hepatitis B virus.Pregnant women whose HBsAg and HBeAg are positive are included in the study.Eligible hepatitis B pregnant women are given TAF antiviral therapy at 24-28 weeks of gestation to block mother-to-child transmission and followed up during pregnancy and after delivery.The study will be initiated with approval by the central ethics committee.Subjects will start screening after signing the informed consent form. Those who meet the criteria will start taking TAF (25mg, oral, 1/day) at 24-28 weeks of gestation until one month after delivery.At that time, chronic hepatitis B carrier will stop taking antiviral therapy, and patients with chronic hepatitis B decide whether to continue the therapy according to the patient's condition.The babies born are immunized according to the national standard immunization program,, that is, 100 IU of hepatitis B immunoglobulin (HBIG) and 10 μg/0.5 ml of hepatitis B vaccine are given within 12 hours after birth. And the same dose of hepatitis B vaccine is given at 1 month and 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* maternal age: 20 to 35 years
* 20-24 week of gestation
* HBsAg-positive more than 6 months and HBeAg-positive
* HBV DNA> 1000,000 IU/ml
* both husband and wife voluntarily sign informed consent
* with good compliance and comply with follow-up programs

Exclusion Criteria:

* mother with co-infection of hepatitis C virus,human immunodeficiency virus
* evidence of decompensated liver disease
* combined with important organ lesions which will affect patient compliance and follow-up plans, pregnant women who are expected to be difficult to complete the study
* have a history of spontaneous abortion, or have a birth defect or congenital malformation in the last pregnancy
* mother treated with antiviral therapy within 6 months prior to enrollment(except those treated with antiviral therapy in the last pregnancy to prevent mother-to-child transmission)
* have a history of kidney injury, creatinine clearance <50ml/min, urine protein positive (>300mg/L)
* combined with other chronic diseases and need to take immunomodulators, cytotoxic drugs or hormonal drugs during pregnancy
* the infants' biologic father is a chronic HBV infected person
* symptoms of threatened abortion during early pregnancy
* evidence of hepatic cell carcinoma
* alanine aminotransferase (ALT) > 10 x upper limit of normal(ULN ), or total bilirubin (TBIL) > 3 x ULN or glomerular filtration rate (GFR) < 90 mL (min*1.73 m2), or serum Albumin (ALB) < 25 g/L before enrollment
* fetal malformations detected by B-ultrasound
* participants in other research

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women in the Affiliated Nanjing Hospital of Nanjing University of Chinese Medicine (The Second Hospital of Nanjing) whose HBsAg and HBeAg are positive are enrolled in the study. TAF is used as antiviral therapy during 24-28 week of gestation.The safety and efficacy of TAF are evaluated.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
MTCT rates in the TAF treated mothers | 28 weeks post-partum
  detectable levels of HBV DNA or HBsAg in the peripheral serum samples of infants at age 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Hospital of Nanjing University of Chinese Medicine (The Second Hospital of Nanjing), Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Han G, Zhou G, Sun T, Luo X, Xu J, Chen C, Xu W, Jiang S, Wang C. Tenofovir alafenamide in blocking mother-to-child transmission of hepatitis B virus: a multi-center, prospective study. J Matern Fetal Neonatal Med. 2022 Dec;35(26):10551-10558. doi: 10.1080/14767058.2022.2134771. Epub 2022 Oct 17. PMID 36253882